CLINICAL TRIAL: NCT03185559
Title: A Prospective, Randomized, Double-blind, Parallel-group, Sham Controlled Single-center Pivotal Clinical Investigation to Evaluate the Clinical Safety and Performance of Self-administered Home-use Combined Occipital and Supraorbital Transcutaneous Nerve Stimulation Device (Relievion™) in Treating Migraine.
Brief Title: A Randomized, Double-blind Clinical Investigation to Evaluate the Use of the Relievion™ Device in Treating Migraine.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator retierment
Sponsor: Neurolief Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NRLF-0038-17-MMC-CTIL
Record Dates: First submitted 2017-06-11; First posted 2017-06-14 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Relievion device- Treatment stimulation (Active Comparator): Relievion Device- Treatment combined occipital and supraorbital transcutaneous nerve stimulation
  Interventions: Device: Relievion Device- Treatment Stimulation
- Relievion device- Sham Stimulation (Sham Comparator): Relievion Device- Sham combined occipital and supraorbital transcutaneous nerve stimulation
  Interventions: Device: Relievion Device- Sham stimulation

INTERVENTIONS:
Device: Relievion Device- Treatment Stimulation — 1 Hour self-administered treatment specific occipital and supraorbital transcutaneous nerve stimulation
  Other Names: Neurolief device
  Arms: Relievion device- Treatment stimulation
Device: Relievion Device- Sham stimulation — 1 Hour self-administered sham occipital and supraorbital transcutaneous nerve stimulation
  Other Names: Sham Neurolief device
  Arms: Relievion device- Sham Stimulation

SUMMARY:
This study will evaluate the clinical performance and safety of a self-administered abortive treatment for migraine headache using combined occipital and supraorbital transcutaneous nerve stimulator (Neurolief device, Relievion™).

ELIGIBILITY:
Inclusion Criteria:

* History of episodic or chronic migraine with or without aura meeting the diagnostic criteria listed in ICHD-III (International Classification of Headache Disorders) beta (2013) section 1, migraine, with the exception of ''complicated migraine'' (i.e., hemiplegic migraine, basilar-type migraine, ophthalmoplegic migraine, migrainous infarction).
* Capable of cooperating with the study protocol and to sign an informed consent.

Exclusion Criteria:

* Patients having received Botox treatment in the head region in the prior 4 months.
* Patients having received supraorbital or occipital nerve blocks in the prior 4 months.
* History of Medication Overuse Headache.
* Patients using opioid medication.
* Allodynia: intolerance to supraorbital and/or occipital neurostimulation (allodynia) that makes the treatment not applicable (the patients will be excluded if they are unable to tolerate the first 3 minutes of neurostimulation).
* Implanted metal or electrical devices in the head (not including dental implants).
* Patient having had a previous experience with the Relievion™ device.
* Patients who have concomitant epilepsy.
* History of neurosurgical interventions.
* Patients with implanted neurostimulators, surgical clips (above the shoulder line) or any medical pumps.
* History of drug abuse or alcoholism.
* Participation in current clinical study or participated in a clinical study within 3 months prior to this study.
* Skin lesion or inflammation at the region of the stimulating electrodes.
* Personality or somatoform disorder.
* Pregnancy or Lactation.
* Women of reproductive age not using efficient contraceptive method.
* History of cerebrovascular event.
* Subjects with recent brain or facial trauma (occurred less than 3 months prior to this study).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-07-23 (Actual); Primary Completion 2018-01-09 (Actual); Study Completion 2018-01-09 (Actual)

PRIMARY OUTCOMES:
Pain Visual Analogue Scale (VAS) Change from basline to 1 hour | 1 Hour
  Mean change of pain score (measured on a visual analog scale) at 1 hour compared to baseline (if rescue therapy was not used)

SECONDARY OUTCOMES:
Pain VAS change from baseline to 30 minutes | 30 minutes
  Mean change of pain score (measured on a visual analog scale) at 30 minutes compared to baseline (if rescue therapy was not used).
Pain VAS change from baseline to 2 hours | 2 Hours
  Mean change of pain score (measured on a visual analog scale) at 2 hours compared to baseline (if rescue therapy was not used).
Pain VAS change from baseline to 24 hours | 24 Hours
  Mean change of pain score (measured on a visual analog scale) at 24 hours compared to baseline (if rescue therapy was not used).
Pain VAS change from baseline to 48 hours | 48 Hours
  Mean change of pain score (measured on a visual analog scale) at 48 hours compared to baseline (if rescue therapy was not used).
Rescue medication at 2 hours | 2 hours
  Proportion of patients not having required rescue medication at 2 hours
Rescue medication within 24 hours | 24 hours
  Proportion of patients not having required rescue medication within 24 hours
Rescue medication within 48 hours | 48 hours
  Proportion of patients not having required rescue medication within 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Colin Klein, Dr, Principal Investigator — Meir Medical Center, Kfar Saba, Israel
Locations (1):
- Meir General Hospital, Kfar Saba, Israel

IPD SHARING:
Plan to Share IPD: No